CLINICAL TRIAL: NCT01386814
Title: Aspects of Neuropsychological Assessment, Standard and Sleep Efficiency in People Exposed to Altitude
Brief Title: Neuropsychological Sleep Physical Exercise Hypoxia
Acronym: Hypoxia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Marco Túlio de Mello, Federal University of São Paulo
Other Study IDs: CEP 1110/08
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-05

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aim: To evaluate the influence of oxygen deficit on the cognitive performance and also about the architecture and sleep efficiency in volunteers subjected to mild and moderate exercise in a hypobaric chamber. SUMMARY: Participants in this study 30 healthy male volunteers, aged 20 to 40 years, regular physical activity, constituting three groups: 1 - without exercise-hypoxia group 10 volunteers who not be subjected to any kind of physical exercise in hypoxia and remain all day of experiment, 2 - group exercise at sea level, is composed of 10 volunteers who will undergo a protocol exercise physical sea-level, 3 - group exercise and hypoxia - 10 volunteers who will carry out a protocol exercise on a treadmill, being the same in condition of hypoxia (hypobaric chamber). All groups on the first day of the experiment will undergo baseline assessments, laboratory blood analysis salivary and spirometric testing. Assessments will be personality and neuropsychological. After baseline assessments, the last day of the experiment, the groups will be evaluated again 4350m above sea level the sea, by personality tests, neuropsychological and laboratory. RATIONALE AND BACKGROUND: During exposure to environments with a partial reduction of oxygen, human body can undergo several physiological and psychological changes are not prepared for such condition. Few studies have reported that the elevation changes and cognitive aspects related to sleep.

MATERIAL AND METHOD: They describe the procedures to be performed, and the study conducted in local with adequate infrastructure.

DETAILED DESCRIPTION:
ADDITIONAL RISKS TO THE PATIENT: Minimal risk, mild discomfort, involving blood collect. Purpose: To evaluate the influence of oxygen deficit on the cognitive performance and also about the architecture and sleep efficiency in volunteers subjected to mild and moderate exercise in a hypobaric chamber.

SUMMARY: Participants in this study 30 healthy male volunteers, aged 20 to 40 years, regular physical activity, constituting three groups: 1 - without exercise-hypoxia group 10 volunteers who not be subjected to any kind of physical exercise in hypoxia and remain all day of experiment, 2 - group exercise at sea level, is composed of 10 volunteers who will undergo a protocol exercise physical sea-level, 3 - group exercise and hypoxia - 10 volunteers who will carry out a protocol exercise on a treadmill, being the same in condition of hypoxia (hypobaric chamber). All groups on the first day of the experiment will undergo baseline assessments, laboratory blood analysis salivary and spirometric testing. Assessments will be personality and neuropsychological. After baseline assessments, the last day of the experiment, the groups will be evaluated again 4350m above sea level the sea, by personality tests, neuropsychological and laboratory. RATIONALE AND BACKGROUND: During exposure to environments with a partial reduction of oxygen, human body can undergo several physiological and psychological changes are not prepared for such condition. Few studies have reported that the elevation changes and cognitive aspects related to sleep

ELIGIBILITY:
Inclusion Criteria:Be physically active (perform aerobic exercise at least three times a week for at least 1 year);

* Minimum age 12 years school;
* Intelligence quotient ≥ 80.

Exclusion Criteria:Present health problems (as assessed by cardiac and respiratory care) and those that do not allow the practice of exercise;

* Present changes in resting electrocardiogram and effort and in clinical evaluation conducted by the Medical Center for Psychobiology and Exercise;
* Being a smoker and / or using drugs of abuse;
* Make use of psychotropic medications;
* Make use of alcoholic beverages frequently;
* Display sleep disorders

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in this study 30 healthy male volunteers, aged 20 to 40 years, regular physical activity, constituting three groups: 1 - without exercise-hypoxia group 10 volunteers who not be subjected to any kind of physical exercise in hypoxia and remain all day of experiment, 2 - group exercise at sea level, is composed of 10 volunteers who will undergo a protocol exercicio physical sea-level, 3 - group exercise and hypoxia - 10 volunteers who will carry out a protocol exercise on a treadmill, being the same in condition of hypoxia. All groups on the first day of the experiment will undergo baseline assessments, laboratory blood analysis salivary and spirometric testing.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marco T Mello, Dr, Principal Investigator — Federal University of São Paulo